CLINICAL TRIAL: NCT01403805
Title: The Interventional Study in the Effects of Oral Care With Vaccines at Nursing Home; the Role of the Partnership With Physician, Dentist and Other Co-medical Stuff
Brief Title: Effects of the Oral Care With Vaccines for Pneumonia in Elderly; Going Home Together Both Physician and Dentist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yubari Kibounomori (Other)
Collaborators: Health Research Foundation (Other)
Responsible Party: Principal Investigator, Masahiro Hatta, Dr., Yubari Kibounomori
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 803121
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Pneumonia
Keywords: Oral care; Vaccine; Pneumonia; Elderly; Prevention; Primary care
MeSH Terms: conditions — Pneumonia | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral care and vaccines (Experimental): Oral care and pneumococcal plus influenza vaccines
  Interventions: Biological: Pneumococcal vaccination (Pneumovax NP, 21800AMY10131000); Biological: Influenza vaccination (Flubik HA, 16100EZZ01207000); Other: Specific frequency of oral care
- Vaccine (Active Comparator): Influenza vaccine only
  Interventions: Biological: Influenza vaccination (Flubik HA, 16100EZZ01207000)

INTERVENTIONS:
Biological: Pneumococcal vaccination (Pneumovax NP, 21800AMY10131000) — Injection,subcutaneous,0.5ml,ones,Planned duration of intervention:a day
  Other Names: Pneumovax NP; Serial Number: 21800AMY10131000
  Arms: Oral care and vaccines
Biological: Influenza vaccination (Flubik HA, 16100EZZ01207000) — Injection,subcutaneous,0.5ml,ones,Planned duration of intervention:a day
  Other Names: Flubik HA; Serial Number: 16100EZZ01207000
  Arms: Oral care and vaccines
Biological: Influenza vaccination (Flubik HA, 16100EZZ01207000) — Injection,subcutaneous,0.5ml,ones,Planned duration of intervention:a day
  Other Names: Flubik HA; Serial Number: 16100EZZ01207000
  Arms: Vaccine
Other: Specific frequency of oral care — 1 dentist and 2 dental hygienists visited the nursing home once a week. After the residents agreed our receive oral care, the dentist/dental hygienist spent 15 minutes with brushing of teeth, scaling, oral wiping, gargling and cleaning of dentures, to reduce dental plaque which is oral bacteria mechanically by using cleaning tools, including toothbrush, interdental brush, dental scaler, tongue brush, and sponge brush to treatment of periodontal disease at the washstand in their private room primary care physicians. At the same time, they taught and recorded to the nursing care workers the methods of administering responsible oral care to dye for dental plaque by using plaque disclosing agent material.
  Other Names: Not applicable:Behaviour
  Arms: Oral care and vaccines

SUMMARY:
Prospective study comparing the effects of interventions (combined oral care and pneumococcal plus influenza vaccinations) in preventing pneumonia and increasing the survival rate from pneumonia.

DETAILED DESCRIPTION:
The elderly population can be expected to increase not only in developed countries, but also in developing countries. Pneumonia is one of the most common causes of death in the elderly.

The investigators conducted a prospective study comparing the effects of interventions (combined oral care and pneumococcal plus influenza vaccinations) in preventing pneumonia and increasing the survival rate from pneumonia in consecutive elderly patients at a nursing home in Yubari during one year from 2009, with the results in a non-intervention group.

ELIGIBILITY:
Inclusion Criteria:

* The residents or an agent who understand the purpose of this study and give informed consent.

Exclusion Criteria:

* The residents contraindicated to vaccine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hirofumi Hashimoto, M.D.,Ph.D., Study Director — Yubari Health Care Research Center; Masahiro Hatta, D.D.S., Study Chair — Yubari Kibounomori; Takahiro Ichiki, M.D., Study Director — Mukawa town National Health Insurance Hobetsu clinic; Katsushi Nagamori, M.D., Study Director — Yubari Health Care Research Center; Hiroyuki Morita, M.D., Principal Investigator — Yubari Health Care Research Cente; Masako Hatta, D.D.S., Study Director — Yubari Health Care Research Center; Tomohiko Murakami, M.D., Study Director — Yubari Kibounomori
Locations (1):
- Yubari Kibounomori, Yūbari, Hokkaido, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Influenza Vaccine: Number of Participants with only an influenza vaccine(Flubik HA, 0.5ml, Mitsubishi Tanabe Pharm. Co.Ltd.).
- Oral Care With Influenza and Pneumococcal Vaccines: Number of Participants with oral care and both an influenza vaccines (Flubik HA, 0.5ml, Mitsubishi Tanabe Pharm. Co.Ltd.) and a pneumococcal vaccine (PNEUMOVAX NP, 0.5ml, MSD Co.Ltd.) How to do oral care is the following;
  1 dentist and 2 dental hygienists visited the nursing home once a week. After the residents agreed our receive oral care, the dentist/dental hygienist spent 15 minutes with brushing of teeth, scaling, oral wiping, gargling and cleaning of dentures, to reduce dental plaque which is oral bacteria mechanically by using cleaning tools, including toothbrush, interdental brush, dental scaler, tongue brush, and sponge brush to treatment of periodontal disease at the washstand in their private room. At the same time, we taught and recorded to the nursing care workers the methods of administering responsible oral care to dye for dental plaque by using plaque disclosing agent material.
Period: Overall Study
Arm/Group | Influenza Vaccine | Oral Care With Influenza and Pneumococcal Vaccines
Started | 94 | 105
Pneumonia Diagnosis | 21 | 2
Completed | 94 | 98
Not Completed | 0 | 7
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine | Oral Care With Influenza and Pneumococcal Vaccines | Total
Number analyzed (Participants) | 94 | 105 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 92 | 105 | 197
Age Continuous [Mean (Standard Deviation); unit: years] | 85.0 (7.48) | 86.0 (7.64) | 85.5 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 77 | 143
  Male | 28 | 28 | 56
Region of Enrollment [Number; unit: participants]
  Japan | 94 | 105 | 199

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pneumonia
Description: Number of Participants with Pneumonia sufferers
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Influenza Vaccine | Oral Care With Influenza and Pneumococcal Vaccines
Number analyzed (Participants) | 94 | 105
participants | 21 | 2
Statistical Analysis 1: Comparison: Influenza Vaccine vs Oral Care With Influenza and Pneumococcal Vaccines; The results were analyzed as means ± standard deviation (SD) or numbers (%). Differences between the 2 nursing homes were compared using Fisher's test; Test type: Superiority or Other; p < 0.001, Fisher Exact — Fisher's test 'Vaccine' versus 'Oral Care and Vaccines' and 'phumonia' and 'not pneumonia'

2. Secondary Outcome: Death From Pneumonia
Description: Number of participants for the death from pneumonia
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Influenza Vaccine | Oral Care With Influenza and Pneumococcal Vaccines
Number analyzed (Participants) | 94 | 105
participants | 8 | 1
Statistical Analysis 1: Comparison: Influenza Vaccine vs Oral Care With Influenza and Pneumococcal Vaccines; The results are expressed as means ± standard deviation (SD) or numbers (%). Differences between the 2 nursing homes were compared using Fisher's test; Test type: Superiority or Other; p = 0.05, Fisher Exact

3. Other Pre Specified Outcome: Leaving Nursing Home
Description: Numer of resident for leaving nursing home
Time Frame: These participants were followed for the duration of nursing home stay, an average of 22 weeks.
Population: These participants were determined as "Not Completed" due to "Leaving nursing home". We excluded these participants from analysis for outcome measure.
Measure: Number; unit: participants
Groups:
- Leaving Nursing Home: Numer of resident for leaving nursing home
Arm/Group | Leaving Nursing Home
Number analyzed (Participants) | 2
participants | 2

4. Other Pre Specified Outcome: Reject Oral Care
Description: Number of resident to reject oral care
Time Frame: This participant rejected oral care before treatment, Day 1
Population: This participant was determined as "Not Completed" due to "Reject oral care". We excluded this participant from analysis for outcome measure.
Measure: Number; unit: participants
Groups:
- Reject Oral Care: Number of resident to reject oral care
Arm/Group | Reject Oral Care
Number analyzed (Participants) | 1
participants | 1

5. Other Pre Specified Outcome: Reject Vaccine
Description: Number of resident to reject vaccine
Time Frame: These participants rejected vaccine before treatment, Day 1
Population: These participants were determined as "Not Completed" due to "Reject vaccine". We excluded these participants from analysis for outcome measure.
Measure: Number; unit: participants
Groups:
- Reject Vaccine: Number of resident to reject vaccine
Arm/Group | Reject Vaccine
Number analyzed (Participants) | 3
participants | 3

6. Other Pre Specified Outcome: Died Before Oral Care Starting
Description: Number of resident died before the start of oral care
Time Frame: This participant was died before treatment, Day 1
Population: This participant was determined as "Not Completed" due to "Died before oral care starting". We excluded this participant from analysis for outcome measure.
Measure: Number; unit: participants
Groups:
- Died Before Oral Care Starting: Number of resident died before the start of oral care
Arm/Group | Died Before Oral Care Starting
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: 1 year
Description: Died in Period from pneumonia
Arm/Group | Influenza Vaccine | Oral Care With Influenza and Pneumococcal Vaccines
Serious Adverse Events (participants affected / at risk) | 8/94 | 2/105
Other Adverse Events (participants affected / at risk) | 0/94 | 0/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza Vaccine (N=94) | Oral Care With Influenza and Pneumococcal Vaccines (N=105)
Died in period (Infections and infestations) | 8 (8) | 1 (1) — 9 (4.5%) of the 199 eligible participants were death from pneumonia still in period.
Died before trial (Infections and infestations) | 0 (0) | 1 (1) — One participant was died before trial.

LIMITATIONS AND CAVEATS:
small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes